CLINICAL TRIAL: NCT02646371
Title: Phase 2b, Double-blind, Placebo-controlled Efficacy Challenge Study With a Candidate Bioconjugate Vaccine Against Shigella Flexneri 2a
Brief Title: Phase 2b Challenge Study With the Bioconjugate Vaccine Flexyn2a
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LimmaTech Biologics AG (Industry)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SF2A-2B
Record Dates: First submitted 2015-12-23; First posted 2016-01-05 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Shigellosis
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flexyn2a (Active Comparator): 2 doses of 10 μg of Flexyn2a will be injected intramuscularly 4 weeks apart
  Interventions: Biological: Flexyn2a
- Placebo (Placebo Comparator): 2 doses of TBS solution will be injected intramuscularly 4 weeks apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Flexyn2a — 2 doses of 10 μg of Flexyn2a will be injected intramuscularly 4 weeks apart
  Arms: Flexyn2a
Biological: Placebo — 2 doses of TBS solution will be injected intramuscularly 4 weeks apart
  Arms: Placebo

SUMMARY:
In this proof of concept challenge study, the bioconjugate candidate vaccine Flexyn2a will be tested for its ability to induce an immune response that protects healthy adult volunteers from infection with a wild-type Shigella flexneri 2a strain compared to subjects receiving placebo.

DETAILED DESCRIPTION:
Flexyn2a is a bioconjugate candidate vaccine that is able to induce an humoral immune response specific for the 2a-antigen of Shigella flexneri 2a bacteria. Healthy adult volunteers naïve for Shigella flexneri 2a infections at screening will receive two administrations of 10 micrograms Flexyn2a or placebo 4 weeks apart. Four weeks after the second vaccination, each subject will be challenged with 1500 cfu of the virulent Shigella flexneri 2a strain 2457T. In order to assess the ability of Flexyn2a to protect against infection with this strain, the attack rate of shigellosis in the group vaccinated with Flexyn2a will be compared to the group of the subjects who received placebo injections.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-50 years (inclusive)
* Good health, without clinically significant medical history or physical examination findings.
* Negative serum pregnancy test at screening, and negative urine before each vaccination and before challenge for female subjects of childbearing potential.
* Females of childbearing potential must agree to avoid pregnancy by use of effective contraception. Abstinence is not acceptable as effective contraception. Female subjects unable to bear children must have this documented (e.g. tubal ligation or hysterectomy).
* Willingness to participate in the study after all aspects of the protocol have been explained and written informed consent obtained.
* Completion of a training session and demonstrated comprehension of the protocol procedures, knowledge of Shigella-associated illness, and a passing score of 70% or better on a written examination.
* Availability for the study duration, including all planned follow-up visits.
* Willingness to refrain from participating in other studies of investigational products until completion of the last study visit.

Exclusion Criteria:

* Women currently nursing.
* Presence of a significant medical or psychiatric condition which in the opinion of the investigator precludes participation in the study.
* Clinically significant abnormalities in screening hematology or serum chemistry as determined by PI or PI in consultation with the research monitor and sponsor.
* Presence in the serum of HIV antibody, HBs-Ag, or HCV antibody (if confirmed positive by HepC confirmatory test, i.e. RIBA, PCR)
* Evidence of IgA deficiency (serum IgA < 7 mg/dl or limit of detection of assay).
* Evidence of current excessive alcohol consumption or drug dependence.
* Evidence of impaired immune function.
* BMI <19 and ≥35
* Recent vaccination or receipt of an investigational product (within 30 days before vaccination and until last study visit).
* Personal history of an inflammatory arthritis.
* Positive blood test for HLA-B27.
* Personal history of irritable bowel syndrome as defined by Rome III criteria.
* Treatment with immunoglobulins or blood products within 3 months from first candidate vaccine injection.
* Regularly abnormal stool pattern (fewer than 3 per week or more than 3 per day) or loose or liquid stools
* Regular use of laxatives, antacids, or other agents to lower stomach acidity.
* Use of any medication known to affect the immune function (e.g., systemic steroids) within 30 days preceding the first vaccination or planned use during the entire study period.
* Known allergy to any of the following antibiotics: ciprofloxacin, trimethoprim-sulfamethoxazole or penicillin.
* Symptoms consistent with Traveler's Diarrhea concurrent with travel to countries where Shigella infection is endemic (most of the developing world) within two years prior to dosing, OR planned travel to endemic countries during the length of the study.
* Vaccination for or ingestion of Shigella within 3 years prior to vaccination.
* Use of antibiotics during the 7 days before vaccination and challenge
* Use of proton pump inhibitors, H2 blockers or antacids within 48 hours prior to challenge.
* Serum IgG titer to Shigella flexneri 2a LPS ≥ 2500
* Current occupation involving handling of Shigella bacteria
* History of allergy to any vaccine or to soy
* Any other criteria which, in the investigator's opinion, would compromise the ability of the subject to participate in the study, the safety of the study, or the results of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar R Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Patricia Martin, PhD, Study Director — LimmaTech Biologics AG
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, CIR, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Talaat KR, Alaimo C, Martin P, Bourgeois AL, Dreyer AM, Kaminski RW, Porter CK, Chakraborty S, Clarkson KA, Brubaker J, Elwood D, Frolich R, DeNearing B, Weerts H, Feijoo BL, Halpern J, Sack D, Riddle MS, Fonck VG. Human challenge study with a Shigella bioconjugate vaccine: Analyses of clinical efficacy and correlate of protection. EBioMedicine. 2021 Apr;66:103310. doi: 10.1016/j.ebiom.2021.103310. Epub 2021 Apr 13. PMID 33862589

RESULTS

PARTICIPANT FLOW:
Groups:
- Flexyn2a - Vaccination: 2 doses of 10 μg of Flexyn2a will be injected intramuscularly 4 weeks apart
  Flexyn2a: 2 doses of 10 μg of Flexyn2a will be injected intramuscularly 4 weeks apart
- Placebo - Vaccination: 2 doses of TBS solution will be injected intramuscularly 4 weeks apart
  Placebo: 2 doses of TBS solution will be injected intramuscularly 4 weeks apart
Period: Overall Study
Arm/Group | Flexyn2a - Vaccination | Placebo - Vaccination
Started | 34 | 33
Completed | 34 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flexyn2a - Vaccination | Placebo - Vaccination | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Full Range); unit: years] | 36.6 [23.5 to 49.8] | 34.4 [22.3 to 50.3] | 35.5 [22.3 to 50.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Attack Rate of Shigellosis in Vaccinated Subjects.
Description: The attack rate of shigellosis after challenge in vaccine group versus in placebo group was analyzed.
Time Frame: Between Day 56 and Day 64
Measure: Count of Participants; unit: Participants
Groups:
- Flexyn2a: The Flexyn2a treatment arm that was challenged.
- Placebo: The control (Placebo) treatment arm that was challenged.
Arm/Group | Flexyn2a | Placebo
Number analyzed (Participants) | 30 | 29
Participants | 13 | 18

ADVERSE EVENTS:
Groups:
- Flexyn2a - Vaccination: In the Flexyn2a treatment arm - 34 subjects received the first Flexyn2a vaccine and 34 subjects received the second Flexyn2a vaccine.
- Placebo - Vaccination: In the control treatment (Placebo) arm - 34 subjects received the first Placebo vaccine and 30 subjects received the second Placebo vaccine.
Arm/Group | Flexyn2a - Vaccination | Placebo - Vaccination
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 18/34 | 13/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flexyn2a - Vaccination (N=34) | Placebo - Vaccination (N=33)
Unsolicited (Blood and lymphatic) (Blood and lymphatic system disorders) | 7 | 4
Unsolicited (Cardiac disorders) (Cardiac disorders) | 1 | 0
Unsolicited (Eye disorders) (Eye disorders) | 1 | 0
Unsolicited (Gastrointestinal disorders) (Gastrointestinal disorders) | 2 | 2
Unsolicited (General disorders and administration site conditions) (General disorders) | 2 | 1
Unsolicited (Infections and infestations) (Infections and infestations) | 3 | 3
Unsolicited (Injury, poisoning and procedural complications) (Injury, poisoning and procedural complications) | 1 | 1
Unsolicited (Investigations) (Investigations) | 6 | 1
Unsolicited (Metabolism and nutrition disorders) (Metabolism and nutrition disorders) | 5 | 1
Unsolicited (Musculoskeletal and connective tissue disorders) (Musculoskeletal and connective tissue disorders) | 3 | 2
Unsolicited (Respiratory, thoracic and mediastinal disorders) (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Unsolicited (Skin and subcutaneous tissue disorders) (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other